CLINICAL TRIAL: NCT03548350
Title: School Based Physical Activity Interventions and Its Impact on Wellbeing and Educational Outcomes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Dr Mark Tully, Academic supervisor, Queen's University, Belfast
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HealthyKidz
Record Dates: First submitted 2018-05-14; First posted 2018-06-07 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Physical Activity; Health Behavior
MeSH Terms: conditions — Motor Activity; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The experimental group will participate in a 24 week multi-component programme that includes four strands:
  * A physical literacy programme focusing on core elements of strength, agility, speed, balance and flexibility. Delivered by external facilitators for one hour per week over 16 weeks of the programme (2 x8week blocks).
  * 'Golden Mile' - pupils and teachers participate 15min walk/run a min of 2 times per week
  * After schools club (not compulsory) featuring mind-set component delivered by external facilitators
  * Healthy kidz app with reward system
  Interventions: Behavioral: HealthyKidz physical activity programme
- Control (No Intervention): The control group will continue doing physical activity including physical education as is normal for their school

INTERVENTIONS:
Behavioral: HealthyKidz physical activity programme — A 24 week physical activity intervention to promote fitness and wellbeing in primary schools
  Arms: Intervention

SUMMARY:
A school based Physical Activity intervention for pupils (8-9 years old) to promote fitness and wellbeing

DETAILED DESCRIPTION:
The experimental group will participate in a 24 week multi-component programme that includes four strands:

* A physical literacy programme focusing on core elements of strength, agility, speed, balance and flexibility. Delivered by external facilitators for one hour per week over 16 weeks of the programme (2 x8week blocks).
* 'Golden Mile' - pupils and teachers participate 15min walk/run a min of 2 times per week
* After schools club (not compulsory) featuring mind-set component delivered by external facilitators
* Healthy kidz app with reward system

The control group will continue doing physical activity including physical education as is normal for their school

All groups will participate in fitness assessments at week 1 and week 24 of the programme and pupils will also complete questionnaires based on measures described above at week 1 and week 24.

ELIGIBILITY:
Inclusion Criteria:

* aged 8-9 years
* enrolled in participating school

Exclusion Criteria:

* Unable to give informed consent
* Presence of an underlying medical conditions
* Already enrolled in a physical activity intervention

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in fitness | Baseline and week 24
  Change from baseline in fitness as assessed as speed and agility (20 second shuttle run), core strength (timed lying leg raise) and flexibility and balance (single standing leg raise).
Change in health related quality of life measured by Kidscreen-10 quality of life and wellbeing in children | Baseline and week 24
  KIDSCREEN is a validated self-report measure of children's subjective health and well-being. Kidscreen-10 is a 10 item instrument which gives a global health related quality of life score. Scores range from 10 to 50, with higher values indicate a higher health related quality of life.
Physical activity behaviour measured by the Physical Activity Questionnaire for Children (PAQ-C) | Week 24
  The Physical Activity Questionnaire for Older Children (PAQ-C) is a validated self-report questionnaire designed to assess moderate to vigorous physical activity in children over a 7 day recall. Items are scored using a 5-point scale and a mean of all 9 items is used to create an overall PAQ-C activity summary score, with higher scores indicating higher levels of physical activity.

SECONDARY OUTCOMES:
Enjoyment of physical activity measured using the Shortened Physical Activity Enjoyment Scale (S-PACES). | Week 24
  Validated scale consisting of seven negatively worded items from the PACES study. Seven items are rated on a 5-point Likert-type type scale ranging from 1 (disagree a lot) to 5 (agree a lot). Items are summed to generate the S-PACES score, and higher scores reflect greater levels of enjoyment.
Self efficacy measured by the Modified Physical Activity Self-Efficacy Scale (PASES) | Week 24
  A validated 8-item measure of self-efficacy using 5 point likert scale for increased sensitivity. The mean score of all eight items is used to indicate the children's PA self-efficacy with lower scores indicating lower self-efficacy.
Social support for physical activity measured by social support sub scale of the Social-Cognitive Measures for Physical Activity | Week 24
  The original scale was based on friend and family only. However, teacher social support scale was devised for the purpose of the study and follows the structure and wording of the family and friends social support for physical activity scales. Each of the 11 items is scored from 1 to 5, where a score of 1 indicates low levels of social support. Scores are summed and then averaged, resulting in a scale mean.
Physical Self-perception measure by the Children's Physical Self-Perception Profile (CY-PSPP) | Week 24
  The CY-PSPP is a 36 item instrument consisting of six scales which represent a hierarchical arrangement of self-worth factors ranging from a global general self-worth scale (GSW) through a global physical self-worth scale (PSW) to four specific physical competence-adequacy sub domains. Item scores for the scale range from 1-4 with the average score being used to represent the value of the scale. Higher values indicate a better self-perception.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Public Health, Queen's University Belfast, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No